CLINICAL TRIAL: NCT05524077
Title: Catheter Ablation Versus Anti-arrhythmic Drugs for Ventricular Tachycardia (CAAD-VT): A Randomised Trial
Brief Title: Catheter Ablation Versus Anti-arrhythmic Drugs for Ventricular Tachycardia
Acronym: CAAD-VT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Saurabh Kumar, Staff Specialist Cardiologist, Western Sydney Local Health District
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAD-VT
Record Dates: First submitted 2022-08-24; First posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Heart Disease Structural Disorder; Ventricular Tachycardia; Cardiomyopathy, Dilated; Sarcoidosis; Cardiomyopathy, Hypertrophic; Cardiomyopathy Ischemic; Cardiomyopathy, Familial; Arrhythmogenic Right Ventricular Cardiomyopathy 1; Arrhythmogenic Left Ventricular Cardiomyopathy
MeSH Terms: conditions — Tachycardia, Ventricular; Cardiomyopathy, Dilated; Sarcoidosis; Cardiomyopathy, Hypertrophic; Cardiomyopathies; Arrhythmogenic Right Ventricular Dysplasia, Familial, 1 | interventions — Anti-Arrhythmia Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Randomisation will be performed using a secure, password-protected web portal (REDCap) and the allocation sequence will be blinded to investigators and participants until the participants have been deemed eligible and enrolled in the study. It will not be possible to maintain blinding after study enrolment because the intervention is invasive.
  Outcome verification will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ablation (Experimental): Patients will be expected to have a catheter ablation procedure within 2 weeks post randomisation and no longer than 30 days post randomisation.
  Medical therapy can be used as a temporising measure before catheter ablation, as is standard of care. If there is breakthrough VT during the period before the clinical procedure, standard practice will be followed in stabilising the ventricular tachycardia (VT) including intravenous short acting anti-arrhythmic drugs (AAD), admission to hospital, internal or external cardioversion. However, preference will be given to scheduling the procedure within 24-48 hours in this situation.
  Interventions: Procedure: Ablation
- Anti-arrhythmic drugs (AAD) (Active Comparator): Patients managed with medical therapy alone by their usual medical practitioners. A protocol aligned with standard clinical care/current clinical guidelines will be provided for guidance, the objective being that the control arm replicates what would constitute standard of care for patients with ventricular tachycardia managed with a non-interventional approach.
  Interventions: Drug: Anti-arrhythmic Drugs (AADs)

INTERVENTIONS:
Procedure: Ablation — Catheter ablation (CA) will be performed in the standard fashion (described in international guidelines for the Management of Patients with Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death from the AHA/ACC/HRS and the expert consensus statement on Catheter Ablation of Ventricular Arrhythmias from HRS/EHRA/APHRS/LAHRS). CA will be performed under conscious sedation or GA by an Electrophysiologist trained in cardiac arrhythmia ablation. CA will be guided by a combination of mapping techniques (standard practice), and described in guidelines for CA for VT. Mapping techniques will include pace, entrainment, activation, and electro-anatomic substrate mapping, where haemodynamically tolerated. Expected procedure duration is 3-6hrs.
  Post-CA, AAD is stopped if patient was drug naïve pre-randomisation. The baseline type/dose of AAD pre-randomisation is continued if the patient was on an AAD pre-randomisation. Repeat ablations are permitted within 30-days post-randomisation.
  Arms: Ablation
Drug: Anti-arrhythmic Drugs (AADs) — Standard care usually encompasses patients who have not previously had AADs, being commenced on sotalol 80mg twice/day. Lower doses may be initiated by treating doctor, as clinically indicated. If there is contraindication to sotalol, another beta-blocker may be initiated using standard doses. Clinicians may consider alternative AADs if there is contraindication to beta-blockers. Doses would be up titrated to the maximal tolerated amount.
  For patients already on an AAD, amiodarone would usually be added, as per VANISH trial.
  They will receive a loading dose 400mg twice/day for 2 weeks, followed by 400mg/day for 4 weeks and 200mg/day thereafter. Patients who have "failed" amiodarone dose <300mg/day will receive a repeat loading dose of 400mg twice/day for 2 weeks, followed by 400mg/day for 1 week, and 300mg/day thereafter.
  If the treating doctor decides to do a CA for VT, the occurrence and timepoint of cross-over will be recorded. Cross-over is estimated to be <2% (VANISH trial).
  Arms: Anti-arrhythmic drugs (AAD)

SUMMARY:
Sudden cardiac death (SCD) due to recurrent ventricular tachycardia (VT) is an important clinical sequela in patients with structural heart disease. VT generally occurs as a result of electrical re-entry in the presence of arrhythmogenic substrate (scar). Scar tissue forms due to an ischemic cardiomyopathy (ICM) from prior coronary obstructive disease or a non-ischemic cardiomyopathy (NICM) from an inflammatory or genetic disease.

AADs can reduce VT recurrence, but have significant limitations in treatment of VT. For example, amiodarone has high rates of side effects/toxicities and a finite effective usage before recurrence. ICDs prevent cardiac arrest and sudden death from VT, but do not stop VT occurring. Recurrent VT and ICD therapies decrease QOL, increase hospital visits, mortality, morbidity and risk of death. Improvement in techniques for mapping and ablation of VT have made CA an alternative.

Currently, there is limited evidence to guide clinicians either toward AAD therapy or CA in patients with NICM. This data shows significant benefit of CA over medical therapy in terms of VT free survival, survival free of VT storm and VT burden. Observational studies suggest that CA is effective in eliminating VT in NICM patients who have failed AADs, resulting in reduction of VT burden and AAD use over long term follow up. Furthermore, there is limited data on the efficacy of CA in early ICM with VT, or advanced ICM with VT. RCT data is almost exclusively on patients with modest ICM with VT, and this is not representative of the real-world scenario of patients with structural heart disease presenting with VT.

Therefore the primary objective is to determine in all patients with structural heart disease and spontaneous or inducible VT, if catheter ablation compared to standard medical therapy with anti-arrhythmic drugs results in a reduction of a composite endpoint of recurrent VT, VT storm and death at a median follow up of 18 months.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for inclusion if they have:

1. ≥1 prior episode of sustained VT in the prior 6 months;

   1. Spontaneous VT: ≥1 episode of monomorphic VT treated by anti-tachycardia pacing (ATP) and/or internal shock by an ICD; lasting ≥30 seconds in the absence of intra-cardiac device therapy that could either be self-terminating or require reversion by pharmacological therapy or external cardioversion;
   2. Spontaneous VT: ≥1 episode of sustained spontaneous monomorphic VT lasting ≥30 seconds documented on Holter, ECG, Loop recorder or other cardiac monitoring device that could either be self-terminating or require reversion by pharmacological therapy or external cardioversion;
   3. Inducible VT: with syncope or palpitations - inducible VT defined as sustained monomorphic VT of CL ≥200 ms lasting for ≥10 s during a cardiac electrophysiology study (note with 4 extrastimuli with or without provocation with isoprenaline);
2. Already a recipient of an implanted cardiac device such as a pacemaker, defibrillator or a cardiac resynchronisation therapy device and/or is indicated to receive one given a new diagnosis of structural heart disease, based on current guideline recommendations;
3. Aged ≥18 years.

Exclusion Criteria:

Patients will be excluded if they are:

1. Unable or unwilling to provide informed consent or patients physician feels there is not significant equipoise to justify randomisation;
2. Women who are pregnant, breast feeding;
3. Medical illness with an anticipated life expectancy <3 months;
4. Unable to complete study procedures or unwilling to be followed up;
5. Have a concomitant illness, physical impairment or mental condition which in the opinion of the study team/ primary care physician could interfere with the conduct of the study including outcome assessments;
6. Known channelopathy such as long QT, short QT, Brugada syndrome, catecholaminergic polymorphic VT;
7. Known prior diagnosis of no structural heart disease, or idiopathic ventricular arrhythmia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite of Recurrent VT or VT storm | Primary outcome will be assessed at 3-, 6-, 12-, 18-, 24-, 30-, 36- months post-randomisation. VT/VT Storm events after the 30-day treatment 'blanking' period after treatment initiation will be included.
  VT (detected by cardiac device as lasting ≥30 seconds or shorter in duration if treated by the ICD).
  VT storm (three or more documented episodes of VT within 24 hours or incessant VT).
Death | Primary outcome will be assessed at 3-, 6-, 12-, 18-, 24-, 30-, 36- months post-randomisation. Death events at any time after randomisation will be included.
  Death (at any time) due to any cause.

SECONDARY OUTCOMES:
Recurrent sustained VT | Outcome will be assessed at 3-, 6-, 12-, 18-, 24-, 30-, 36- months post-randomisation. VT events will be included after the 30-day treatment 'blanking' period after treatment initiation.
  Recurrent sustained VT detected by implanted cardioverter defibrillator (ICD) (VT identified and treated by the ICD with anti-tachycardia pacing (ATP) and/or internal ICD delivered shock or ≥30 seconds of VT if untreated by ICD)
VT storm | Outcome will be assessed at 3-, 6-, 12-, 18-, 24-, 30-, 36- months post-randomisation. VT storm events will be included after the 30-day treatment 'blanking' period after treatment initiation.
  Three or more documented episodes of VT within 24 hours or incessant VT
VT burden | 6 months after randomisation, with a 30-day treatment 'blanking' period after treatment initiation; and 6 months before randomisation
  VT burden (number of episodes of VT in the preceding 6 months compared to the 6 months after randomisation and therapy)
Cardiovascular hospitalisation | Outcome will be assessed at 3-, 6-, 12-, 18-, 24-, 30-, 36- months post-randomisation. Events will be included after the 30-day treatment 'blanking' period after treatment initiation.
  All cardiovascular hospitalisation; heart failure; hospitalisation for arrhythmia
Mortality | Outcome will be assessed at 3-, 6-, 12-, 18-, 24-, 30-, 36- months post-randomisation. Events will be included at any time after randomisation.
  All-cause mortality; cardiovascular mortality; non-cardiac death
Effect of intervention on ventricular function | Outcome will be assessed at 3-, 6-, 12-, 18-, 24-, 30-, 36- months post-randomisation. Events will be included after the 30-day treatment 'blanking' period after treatment initiation.
  Effect of intervention on ventricular function as assessed by transthoracic echocardiography from baseline to 6-, 12-, 24- and 36-months' post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Saurabh Kumar, MBBS, PhD, Principal Investigator — Western Sydney Local Health District
Locations (12):
- Australia (12):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Blacktown Hospital, Blacktown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: No